CLINICAL TRIAL: NCT01447836
Title: Prognostic Value of Indocyanine Clearance Rate for Sepsis Patients in ICU
Brief Title: Indocyanine Clearance Rate and Septic Liver Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guanqing Sun, Resident doctor, Sun Yat-sen University
Other Study IDs: SLICG; 2011180 (Other: The First Affiliated Hospital, Sun Yat-sen University)
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Sepsis
Keywords: indocyanine green; sepsis; liver injury; abdominal perfusion pressure
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for transaminase, hemoglobin, prothrombin time, lactate and oxygen pressure test.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Sepsis patients who are admitted to SICU of our clinical center.
- Control: Postoperative patients who underwent abdominal surgery and then was directly transferred to SICU of our clinical center.

SUMMARY:
Liver injury is a complication of sepsis and septic liver injury has adverse impact upon the outcome. As a measurement for liver function, Plasma clearance rate of indocyanine green (PDR-ICG) always decreased during the early phase of sepsis. So the investigators hypotheses include: PDR-ICG is lower in sepsis patients than non-septic patients in ICU; PDR-ICG may be lower in abdominal sepsis patients than non-abdominal sepsis patients in ICU; PDR-ICG correlates with abdominal perfusion pressure; change of PDR-ICG in early phase correlates with change of transaminase or bilirubin in late phase of sepsis.

DETAILED DESCRIPTION:
Liver injury is a complication of sepsis and septic liver injury has adverse impact upon the outcome. However, changes of transaminase or bilirubin are always not significant during the early phase of sepsis. As another sort of measurement of liver function, plasma clearance rate of indocyanine green (PDR-ICG) always decreased during the early phase of sepsis. So the investigators hypotheses include: PDR-ICG may be lower in sepsis patients than non-septic patients in ICU; PDR-ICG may be lower in abdominal sepsis patients than non-abdominal sepsis patients in ICU; PDR-ICG correlates with abdominal perfusion pressure; change of PDR-ICG in early phase may correlate with change of transaminase or bilirubin in late phase of sepsis. Through this study we also plan to calculate the range of abdominal perfusion pressure that can maintain normal PDR-ICG and the range of PDR-ICG that can maintain normal transaminase or bilirubin level in sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* For control group: the patient does not match the diagnosis criteria of sepsis before the operation; the operation was done in peritoneal cavity; the patient is transferred to SICU directly from surgical room or recovery room; the patient is anticipated to stay in SICU for more than 48 hours.
* For study group: the patient matches the diagnosis criteria of sepsis; the patient is anticipated to stay in SICU for more than 48 hours.

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* The infection is purely caused by virus
* Obstruction of biliary tract, or acute cholangitis, or acute liver abscess, or active hepatitis, or hyperacute/acute liver rejection occurs during study period
* Hemorrhagic shock occurs during study period
* Asthma occurs during study period
* Acute coronary syndrome occurs during study period
* Continuing peripheral circulation dysfunction leads to refractory "low quality" during PDR-ICG measurement
* Comorbidity of the bladder leads to impossibility to measure intra-abdominal pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to SICU of our clinical center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Plasma clearance of indocyanine green | D0, D1, D2

SECONDARY OUTCOMES:
Transaminase | D0, D1, D2, D4, D6
Bilirubin | D0, D1, D2, D4, D6
Prothrombin time | D0, D1, D2, D4, D6
Lactate | D0, D1, D2, D4, D6
γ-glutamyl transpeptidase | D0, D1, D2, D4, D6
Cholinesterase | D0, D1, D2, D4, D6

CONTACTS AND LOCATIONS:
Overall Officials: Guanxiang Dong, MD, PhD, Study Chair — Surgical Intensive Care Unit, The First Affiliated Hospital, Sun Yat-sen University; Guanqing Sun, MD, Principal Investigator — Surgical Intensive Care Unit, The First Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Surgical Intensive Care Unit, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Rank N, Michel C, Haertel C, Lenhart A, Welte M, Meier-Hellmann A, Spies C. N-acetylcysteine increases liver blood flow and improves liver function in septic shock patients: results of a prospective, randomized, double-blind study. Crit Care Med. 2000 Dec;28(12):3799-807. doi: 10.1097/00003246-200012000-00006. PMID 11153617
- [Background] Sakka SG, Reinhart K, Meier-Hellmann A. Does the optimization of cardiac output by fluid loading increase splanchnic blood flow? Br J Anaesth. 2001 May;86(5):657-62. doi: 10.1093/bja/86.5.657. PMID 11575341
- [Background] Poeze M, Ramsay G, Buurman WA, Greve JW, Dentener M, Takala J. Increased hepatosplanchnic inflammation precedes the development of organ dysfunction after elective high-risk surgery. Shock. 2002 Jun;17(6):451-8. doi: 10.1097/00024382-200206000-00002. PMID 12069179
- [Background] Mizushima Y, Tohira H, Mizobata Y, Matsuoka T, Yokota J. Assessment of effective hepatic blood flow in critically ill patients by noninvasive pulse dye-densitometry. Surg Today. 2003;33(2):101-5. doi: 10.1007/s005950300021. PMID 12616369
- [Background] Inal MT, Memis D, Kargi M, Sut N. Prognostic value of indocyanine green elimination assessed with LiMON in septic patients. J Crit Care. 2009 Sep;24(3):329-34. doi: 10.1016/j.jcrc.2008.11.012. Epub 2009 Feb 12. PMID 19327336
- [Background] Kopterides P, Siempos II, Tsangaris I, Tsantes A, Armaganidis A. Procalcitonin-guided algorithms of antibiotic therapy in the intensive care unit: a systematic review and meta-analysis of randomized controlled trials. Crit Care Med. 2010 Nov;38(11):2229-41. doi: 10.1097/CCM.0b013e3181f17bf9. PMID 20729729
- [Background] Kortgen A, Paxian M, Werth M, Recknagel P, Rauchfuss F, Lupp A, Krenn CG, Muller D, Claus RA, Reinhart K, Settmacher U, Bauer M. Prospective assessment of hepatic function and mechanisms of dysfunction in the critically ill. Shock. 2009 Oct;32(4):358-65. doi: 10.1097/SHK.0b013e31819d8204. PMID 19197231
- [Background] Slotman GJ, Fisher CJ Jr, Bone RC, Clemmer TP, Metz CA. Detrimental effects of high-dose methylprednisolone sodium succinate on serum concentrations of hepatic and renal function indicators in severe sepsis and septic shock. The Methylprednisolone Severe Sepsis Study Group. Crit Care Med. 1993 Feb;21(2):191-5. doi: 10.1097/00003246-199302000-00008. PMID 8428468
- [Background] Seibel A, Sakka SG. [Indocyanine green plasma disappearance rate: estimation of abdominal perfusion disturbances]. Anaesthesist. 2010 Dec;59(12):1091-8. doi: 10.1007/s00101-010-1754-2. Epub 2010 Aug 18. German. PMID 20714702
- [Background] Mathes AM, Kubulus D, Weiler J, Bentley A, Waibel L, Wolf B, Bauer I, Rensing H. Melatonin receptors mediate improvements of liver function but not of hepatic perfusion and integrity after hemorrhagic shock in rats. Crit Care Med. 2008 Jan;36(1):24-9. doi: 10.1097/01.CCM.0000292088.33318.F0. PMID 18090374